CLINICAL TRIAL: NCT05710198
Title: A Phase III Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group Trial of the Efficacy of Citicoline Eye Drops 2% on Visual Field Preservation in Patients With Open Angle Glaucoma
Brief Title: Efficacy of Citicoline Eye Drops 2% on Visual Field Preservation in Patients With Open Angle Glaucoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Omikron Italia S.r.l. (Industry)
Collaborators: OPIS Spain (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OMK1P3
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Glaucoma, Open-Angle
Keywords: Glaucoma; Citicoline; Visual field; Open-Angle glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Intervention Model Description: Multicenter, double-blind, randomized, placebo-controlled, parallel-group trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- citicoline eye drops 2% (Experimental): Citicoline eye drops 2%. One drop in the study eye three times daily throughout the 3-year trial. Patients will be treated with any IOP-lowering agent to control IOP and study treatments should be administered at least 20 minutes after IOP lowering medication.
  Interventions: Drug: Citicoline eye drops 2%
- Placebo eye drops (Placebo Comparator): Placebo eye drops. One drop in the study eye three times daily throughout the 3-year trial. Patients will be treated with any IOP-lowering agent to control IOP and study treatments should be administered at least 20 minutes after IOP lowering medication
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Citicoline eye drops 2% — Eye drops containing Citicoline 2%
  Arms: citicoline eye drops 2%
Drug: Placebo — Eye drops containing placebo matching product
  Arms: Placebo eye drops

SUMMARY:
To evaluate the efficacy of citicoline eye drops 2% in reducing visual field deterioration in patients with progressing OAG treated according to best clinical practice. Secondary objectives are assessing the effect of citicoline eye drops 2% on changes in structural parameters measured by Spectral Domain Optical Coherence Tomography (SD-OCT) and evaluating the safety of citicoline eye drops 2%

DETAILED DESCRIPTION:
Background: Primary open angle glaucoma (OAG) is a chronic progressive neurodegenerative disease where intraocular pressure (IOP) is the main and successfully treatable risk factor. Although the treatment effect is quite large, a significant proportion of patients show disease progression with apparently well controlled IOP. Given the similarities with other neurodegenerative diseases - particularly in the mechanisms of cell death - neuroprotective treatments have been tested also in glaucoma. Interesting results from experimental studies and first evidence from human glaucoma trials have been published in recent years.

Citicoline is one of the promising molecules with a putative neuroprotective action and has been evaluated in patients with various neurodegenerative diseases with encouraging results. The mechanism of action of citicoline is multifarious and includes preservation of cardiolipin and sphingomyelin, restoration of phosphatidylcholine, stimulation of glutathione synthesis, lowering of glutamate concentration, rescuing mitochondrial function, and others. Pilot studies on glaucomatous patients showed a possible effect of citicoline as additive therapy in the treatment of glaucoma, in reducing progression of visual field changes, in protecting retinal nerve fiber layers and in improving vision related Quality of Life (QoL), though these findings are yet to be confirmed by a large randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Age ≥ 18 years.
3. Eyes with OAG, Pseudoexfoliation and pigmentary glaucoma will be included.
4. Best Corrected Visual Acuity (BCVA) ≥ 0.5 for the study eye.
5. Controlled IOP (≤ 18 mmHg, average of the last 3 measurements in the clinic) in the study eye.
6. Visual field MD not worse than -12 dB at the latest assessment in the clinic for the study eye.
7. Deteriorating MD at a rate between -0.5 dB/year and -1.0 dB/year, estimated from the latest VF tests collected in the clinic (at least 4) over a period during which incisional glaucoma surgery was not performed. Combinations of SITA Standard and Fast strategies (but not SITA Faster) is admissible. Patients who reach the desired minimum number of tests (4) with a mixture of SITA Standard/Fast and SITA Faster tests will need to perform additional replacement tests according to the prevalent strategy used in their series of VF (i.e. additional SITA Standard/Fast tests if ≤ 2 tests were SITA Faster; additional SITA Faster if > 2 tests were SITA Faster).
8. Glaucoma definition will be based on VF damage (24-2, any SITA strategy) and spatially congruent glaucomatous changes at the ONH. If both eyes are eligible, the eye with the better MD will be chosen as the study eye.
9. Women of childbearing potential willing to use an appropriate method of contraception.

Exclusion Criteria:

1. Cataract in the study eye which, in the opinion of the clinician, may require cataract surgery within the next three years.
2. Only-eye patients (visual acuity < 0.1 decimals in one eye or more than two paracentral VF locations with a sensitivity of < 10 dB).
3. Known intolerance or allergy to any of the components in the eye drops.
4. Diode laser treatment or glaucoma surgery in the past 2 years or cataract surgery within the last 6 months in the study eye.
5. Eyes with any type of glaucoma other than primary, pseudoexfoliative or pigmentary OAG.
6. Patients with other ocular or systemic comorbidities that, in the opinion of the Investigator, might affect the VF or the execution of the test.
7. Patients already on topical or systemic citicoline treatment.
8. Patients taking other systemic or topical potential neuroprotectors competing with citicoline eye drops 2% (a list will be provided) unwilling to suspend these treatments and undergo a washout period of 6 months prior to the study.
9. Patients unable to perform reliable VF tests, based on the assessment of the last 4 available 24-2 Humphrey Field Analyzer (HFA) VF tests performed in the clinic with a false positive rate (FP) ≤ 15%.
10. Pregnant and nursing patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression of visual field damage | 3 years
  Difference in the rate of progression of VF damage in the study eye between the two trial arms. This will be measured with repeated, planned visual field (VF) tests, all performed with a Humphrey Field Analyser (HFA, Zeiss Meditec, Dublin, CA) with the SITA Standard 24-2 strategy, over the span of three years.

SECONDARY OUTCOMES:
Rate of progression in structural parameters | 3 years
  Difference in the rate of progression in structural parameters. These parameters focus on the ocular structures mostly damaged by glaucoma. The parameters of interest will be:
  * RNFL thickness measured with Optical Coherence Tomography (OCT).
  * Inner retina thickness in the macula (RNFL, Ganglion Cell Layer and Ganglion Cell + Inner Plexiform Layer complex).
Safety (IOP) | 3 years
  Safety will be assured by regular assessments of adverse events and IOP. IOP will be carefully monitored and managed as per standard clinical practice (detailed management of IOP is reported later). Side effects from the neuroprotective drops or any IOP lowering treatment, including allergic reactions, ocular surface toxicity and signs of extraocular or intraocular inflammation, will be carefully assessed by the examiners and reported in the case report form (CRF). Any significant discomfort or adverse reactions to the drops or clear signs of inflammation will be reasons for early withdrawal
Visual Field recovery | 3 years
  Evidence of neuro-recovery. The Visual field Mean Deviation values (2 tests) at Visit 2 will be compared between the two groups, after adjusting for the MD values at Visit 1 (baseline, 2 tests).

CONTACTS AND LOCATIONS:
Locations (1):
- Presidio Ospedale San Paolo, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cavaterra D, Giammaria S, Pandino I, Zingale GA, Delli Paoli V, Fiore R, Michelessi M, Roberti G, Carnevale C, Tanga L, Cazzato D, Peroni E, Grasso G, Manni G, Bocedi A, Oddone F, Coletta M, Sbardella D, Tundo GR. Citicoline Triggers Proteome Remodeling and Proteostatic Adaptation: Evidence from Shotgun Proteomics. Pharmaceutics. 2026 Jan 1;18(1):61. doi: 10.3390/pharmaceutics18010061. PMID 41599168